CLINICAL TRIAL: NCT02192593
Title: Randomized Controlled Trial of Computerized Cognitive Behavioral Therapy for Auditory Hallucinations in Persons With Psychosis
Brief Title: Computerized Cognitive-Behavioral Therapy for Auditory Hallucinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Jennifer Gottlieb, Research Assistant Professor, Boston University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ComputerCBTPsychosis
Record Dates: First submitted 2013-09-13; First posted 2014-07-17 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2015-07

CONDITIONS: Schizophrenia, Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer CBT (Experimental): A 10-session computerized cognitive-behavioral therapy intervention
  Interventions: Behavioral: Computer CBT
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Computer CBT
  Arms: Computer CBT

SUMMARY:
This is a randomized controlled trial, examining the effects of a computerized, internet-based Cognitive Behavioral Therapy (CBT) Intervention for persons with a schizophrenia spectrum disorder who experience distressing auditory hallucinations (voices). Participants are randomized to one of two conditions: either to receive the 10-session computer-based program on a weekly basis, or to their usual care at their mental health clinic. This study takes place at Cambridge Health Alliance in Cambridge Massachusetts. It is hypothesized that the participants who participate in the CBT program will have significant improvements in the severity of their auditory hallucinations, as well as their associated distress, compared to the participants receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be on a stable dose of antipsychotic medication for the past 3 months.

  * Schizophrenia-spectrum diagnosis, including schizophrenia, schizoaffective disorder, schizophreniform disorder, and psychosis, not otherwise specified.
  * At least moderate severity on Brief Psychiatric Rating Scale (BPRS) hallucinations item.
  * Naïve to CBTp for Auditory Hallucinations within the past 3 years.
  * No current suicidal ideation or hospitalization within the past month.
  * Reading level of at least 4th grade, as measured by the reading section of the Wide Range Achievement Test (WRAT)
  * Current patient receiving care at Cambridge Health Alliance

Exclusion Criteria:

* Terminal physical illness expected to result in the death of the study participant within one year.

  * Primary diagnosis of dementia or a diagnosis of a psychiatric disorder secondary to a medical condition.
  * Comorbid dementia (severe cognitive impairment) as indicated by a Mini-mental state examination score <24.
  * Current active substance abuse or dependence with the need for specialized substance abuse services
  * Does not speak English
  * Does not achieve a 4th grade reading level as demonstrated on the Wide Range Achievement Test (WRAT)
  * Has a legal guardian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | Baseline, Post-Treatment, 3-Month Follow-up
  Primary outcome is change in BPRS hallucinations item from baseline to post-treatment to 3 month follow-up. This measure assesses severity of auditory hallucinations as well as overall psychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Gottlieb, PhD, Principal Investigator — Boston University
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States